CLINICAL TRIAL: NCT03162575
Title: The Possible Beneficial Effects of Mindfulness-Based Cognitive Therapy (MBCT) in Fatigued Adult Patients With Inflammatory Bowel Disease (IBD)
Brief Title: Mindfulness-Based Cognitive Therapy for Fatigue in Inflammatory Bowel Disease Patients: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maya Schroevers, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016.316
Record Dates: First submitted 2017-05-01; First posted 2017-05-22 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Psychological
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (Experimental): The intervention consists of 8 weekly sessions of MBCT. Each session will be administered in a group and will last 2.5 hours
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Waiting List Control (No Intervention): Patients assigned to the waiting list condition will receive no intervention for three months and afterwards will receive MBCT

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — Structured MBCT intervention based on the protocol of Williams, Teasdale, and Segal (2002)
  Other Names: MBCT
  Arms: Mindfulness-Based Cognitive Therapy

SUMMARY:
The current study aims to investigate the efficacy of Mindfulness-Based Cognitive Therapy (MBCT) for reducing fatigue in Inflammatory Bowel Disease patients in remission.

DETAILED DESCRIPTION:
Fatigue is highly prevalent in patients with inflammatory bowel disease (IBD, i.e. Crohn's disease and ulcerative colitis), and may negatively impact patients' illness management, treatment adherence, and quality of life. Given this burden, effective treatment for reducing fatigue in IBD patients is warranted. A promising psychological treatment is Mindfulness-Based Cognitive Therapy (MBCT). MBCT is a standardized, highly structured eight-week group program for reducing stress, depression, fatigue and/or pain. Several meta-analyses have demonstrated the effectiveness of MBCT in reducing psychological complaints and improving quality of life. Moreover, in patients with cancer or chronic fatigue syndrome, there is preliminary evidence that MBCT can be effective in reducing fatigue. Given this lack of evidence for the efficacy of MBCT in reducing fatigue in general and the specific and strongly illness-related nature of fatigue in patients with IBD and characteristics of the illness, including its lifelong and relapsing nature, there is a need to verify whether MBCT is effective in reducing fatigue in IBD patients with severe fatigue.

This randomized controlled trial (RCT) aims to investigate the efficacy of Mindfulness-Based Cognitive Therapy (MBCT) in reducing fatigue in severely fatigued IBD patients. Additionally, the effects of MBCT on clinically relevant secondary outcomes will be examined: fatigue interference, mood, IBD-specific quality of life, sleep quality, labor participation. Also patients' satisfaction will be assessed. Moreover, mediators and moderators will be examined to increase the understanding of why and for whom MBCT is particularly effective.

A randomized controlled trial will be performed, including two conditions: MBCT and a waitlist control group (who will receive MBCT after a waiting period of three months). The study sample will consist of 128 adult patients with IBD in remission and experiencing severe fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either Crohn's disease or Ulcerative Colitis
* Currently in remission
* No expectation of a surgery in the upcoming three months
* Score on the subscale 'subjective fatigue' of the CIS (8 items) ≥ 35 (i.e. indicating severe fatigue)
* Age ≥ 18 and ≤ 75 years at the time of study entrance
* Being able to attend eight weekly group sessions of 2.5 hours in the hospital
* Being able to read, write, and speak Dutch.
* Written informed consent

Exclusion Criteria:

* Severe cognitive, neurological or psychiatric co-morbidity that could interfere with patients' participation and/or warrant other treatment, including acute suicidal ideations or behavior, diagnosis of schizophrenia or history of psychotic complaints, bipolar disorder, severe personality disorder, or history of clinically significant drug abuse or substance dependence
* Pregnancy
* Anemia (i.e. Hb < 7.4 for women, < 8.1 for men)
* Change in IBD medication (i.e. use of steroids) within 1 month before study entry
* Currently receiving psychological treatment for fatigue or for psychological/psychiatric problems.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
Change in fatigue | Change from baseline in severity of fatigue symptoms at 3 months, 6 months and 12 months
  Fatigue will be assessed with the Checklist Individual Strength (CIS-20)

SECONDARY OUTCOMES:
Change in fatigue interference | Change from baseline in fatigue interference at 3 months, 6 months, and 12 months
  Fatigue interference will be measured by the Fatigue Symptom Inventory (FSI)
Change in anxiety | Change from baseline in generalized anxiety at 3 months, 6 months, and 12 months
  Anxiety will be measured by Generalised Anxiety Disorder Assessment (GAD 7)
Change in depression | Change from baseline in depression at 3 months, 6 months, and 12 months
  Depression will be measured by Beck Depression Inventory-II (BDI-II)
Change in IBD-specific quality of life | Change from baseline in quality of life at 3 months, 6 months, and 12 months
  IBD-specific quality of life will be measured by the IBD-Q
Change in sleep quality | Change from baseline in sleep quality at 3 months, 6 months, and 12 months
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index
Change in labor participation | Change from baseline in labor participation at 3 months, 6 months, and 12 months
  Labor participation will be assessed with several questions
Satisfaction with treatment | Assessed at 3 months
  Satisfaction with treatment will be assessed with several questions

CONTACTS AND LOCATIONS:
Overall Officials: Maya Schroevers, PhD, Principal Investigator — Department of Health Sciences; Gerard Dijkstra, Prof., Principal Investigator — Center for Liver, Digestive and Metabolic Diseases (CLDM)
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Bredero QM, Fleer J, Smink A, Kuiken G, Potjewijd J, Laroy M, Visschedijk MC, Russel M, van der Lugt M, Meijssen MAC, van der Wouden EJ, Dijkstra G, Schroevers MJ. Long-term treatment outcomes of mindfulness-based cognitive therapy for fatigue in patients with inflammatory bowel disease: Results of a randomized controlled trial. J Psychosom Res. 2024 Dec;187:111949. doi: 10.1016/j.jpsychores.2024.111949. Epub 2024 Oct 11. PMID 39418854